CLINICAL TRIAL: NCT00585312
Title: A Phase III Placebo-Controlled Trial Of Celecoxib In Genotype Positive Subjects With Familial Adenomatous Polyposis
Brief Title: Trial In Pediatric Patients With Familial Adenomatous Polyposis (FAP)
Acronym: CHIP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: A3191193; NCT00393016 (obsolete NCT alias); NCT00534040 (obsolete NCT alias)
Record Dates: First submitted 2008-01-01; First posted 2008-01-03 (Estimated); Results first posted 2014-11-03 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Adenomatous Polyposis Coli
Keywords: FAP
MeSH Terms: conditions — Adenomatous Polyposis Coli | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Celecoxib (Experimental): celecoxib, 16 mg/kg/day, for 5 years
  Interventions: Drug: Celecoxib
- Placebo (Placebo Comparator): Masked, placebo comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Celecoxib — celecoxib, 16 mg/kg/day, for 5 years
  Other Names: celebrex, SC-58635
  Arms: Celecoxib
Drug: Placebo — Masked, placebo comparator
  Arms: Placebo

SUMMARY:
To test whether celecoxib can be used to prevent colon polyp formation in children with familial adenomatous polyposis (FAP).

DETAILED DESCRIPTION:
Per DMC recommendation, the study was terminated early (31Oct2013) due to low enrollment and low endpoint accumulation rate. No safety concerns were involved in the decision to terminate the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 10-17 years
* Confirmed deleterious FAP genotype based on central genetic testing or personal history ot >2 colorectal adenomas and a parent with the diagnosis of FAP and either A, B or C below A: Non-attenuated FAP genotype B: Attenuated FAP genotype and a personal history of colorectal adenomas and a first degree relative with FAP C: No genotype identified with a personal history of > 2 adenomas and have a parent with FAP
* Less than 30 polyps, which need to be removed to render the colon polyp-free before study drug can be given

Exclusion Criteria:

* Diagnosis of attenuated FAP based on central genetic testing in the absence of a personal history of >2 colorectal adenomas and a first degree relative (parent or sibling) with FAP.
* Sensitivity to COX-2 inhibitors

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2006-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (38):
- United States (19):
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Chagrin Falls, Ohio
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Elyria, Ohio
  - Pfizer Investigational Site, Independence, Ohio
  - Pfizer Investigational Site, Lakewood, Ohio
  - Pfizer Investigational Site, Lorain, Ohio
  - Pfizer Investigational Site, Solon, Ohio
  - Pfizer Investigational Site, Strongsville, Ohio
  - Pfizer Investigational Site, Westlake, Ohio
  - Pfizer Investigational Site, Willoughby Hills, Ohio
  - Pfizer Investigational Site, Wooster, Ohio
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
- Belgium (2):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Ghent
- Pfizer Investigational Site, Prague, Czechia
- Hong Kong (2):
  - Pfizer Investigational Site, Shatin, New Territories
  - Pfizer Investigational Site, Hong Kong
- Pfizer Investigational Site, Miskolc, Hungary
- Israel (4):
  - Pfizer Investigational Site, Haifa
  - Pfizer Investigational Site, M.P. Lower Galilee
  - Pfizer Investigational Site, Petach Tikvah 49202
  - Pfizer Investigational Site, Tel Aviv
- Italy (2):
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, Siena
- Pfizer Investigational Site, Rio Piedras, Puerto Rico
- Pfizer Investigational Site, Bratislava, Slovakia
- Pfizer Investigational Site, Cape Town, Western Cape, South Africa, South Africa
- Pfizer Investigational Site, Madrid, Spain
- Pfizer Investigational Site, Stockholm, Sweden
- Pfizer Investigational Site, Donetsk, Ukraine
- Pfizer Investigational Site, Harrow, Middlesex, England, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191193&StudyName=Trial%20In%20Pediatric%20Patients%20With%20Familial%20Adenomatous%20Polyposis%20%28FAP%29%0A

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 305 participants were screened, whereof 106 were randomized into the study, and of whom 101 took at least 1 dose of study drug. The clinical study was conducted in 18 centers across 13 countries: Belgium, Czech Republic, Hong Kong, Hungary, Israel, Italy, Slovakia, South Africa, Spain, Sweden, Ukraine, United Kingdom, and United States.
Pre-assignment Details: The randomization was to be stratified by center, age (≥12 years old versus <12 years old), and familial adenomatous polyposis (FAP) phenotype (negative versus positive). The participants were randomized 1:1 to one of the 2 treatments celecoxib or placebo.
Groups:
- Celecoxib: Celecoxib, approximately 16 mg/kg/day (adjusted for changes in body weight). Maximum dose was 400 mg twice daily.
- Placebo: Matching placebo
Period: Overall Study
Arm/Group | Celecoxib | Placebo
Started | 55 (STARTED=Randomized) | 51 (STARTED=Randomized)
Treated | 53 | 48
Completed | 4 | 7
Not Completed | 51 | 44
Not completed — Adverse Event | 3 | 0
Not completed — Lack of Efficacy | 6 | 11
Not completed — Lost to Follow-up | 1 | 1
Not completed — Reason not specified | 2 | 0
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Study terminated by the sponsor | 34 | 31

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population (N: 106) consisted of all participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether the participants received any study drug or received a different drug from that to which they were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Celecoxib | Placebo | Total
Number analyzed (Participants) | 55 | 51 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.6 (2.2) | 12.2 (1.8) | 12.4 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 28 | 57
  Male | 26 | 23 | 49

OUTCOME MEASURES:

1. Primary Outcome: Time to Disease Progression
Description: Time to disease progression was defined as the time from randomization to the earliest occurrence of one or more of the following events:
  1. Appearance of ≥20 polyps (>2 mm in size) at any colonoscopy during the study (Polyps); or
  2. Diagnosis of colorectal malignancy (ColMal).
Time Frame: 5 years
Population: ITT population (N: 106) consisted of all participants who were randomized and assigned to treatment. Primary outcome measure was met by 7 (Polyp:7,ColMal:0) participants in the Celecoxib group and 13 (13,0) in the placebo group. Study was early terminated due to low enrollment and lower than expected endpoint rate. No analysis was performed.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 7 | 13
years | 2.2 (1.08) | 1.8 (1.30)

2. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure was defined as time from randomization to the earliest occurrence of one or more of the following:
  * Appearance of ≥20 polyps (>2 mm in size) at any colonoscopy during the study (Polyps), or
  * Diagnosis of colorectal malignancy (ColMal), or
  * Treatment related dropout (DO). The treatment related dropout was defined as insufficient clinical response, progression of disease, death, adverse event, treatment-related laboratory abnormality, subject no longer willing to participate in study, and other reasons that might be related to treatment as determined by treating physicians in a blind fashion before database release.
Time Frame: 5 years
Population: ITT population (N: 106) consisted of all participants who were randomized and assigned to treatment. Secondary outcome measure was met by 14 (Polyp:7,ColMal:0,DO:14) participants in the Celecoxib and 14 (13,0,12) in the placebo group. Study was early terminated due to low enrollment and lower than expected endpoint rate. No analysis was performed.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 14 | 14
years | 2.0 (1.12) | 1.7 (1.30)

3. Secondary Outcome: Total Number of Colorectal Polyps
Description: Total number of colorectal polyps >2 mm in size, that were detected over Years 1 - 5 cumulatively.
  Weighted total number of colorectal polyps over Years 1 - 5 cumulatively was defined as the total number of colorectal polyps >2 mm in size, that were detected over Years 1 - 5, divided by the number of colonoscopies that the participant had during the study.
Time Frame: Years 1 - 5
Population: ITT population (N: 106) consisted of all participants who were randomized and assigned to a treatment. Study was early terminated due to low enrollment and lower than expected endpoint rate and no analysis was performed.
Measure: Mean (Standard Deviation); unit: polyps
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 55 | 51
polyps
  Year 1 (N: 27, 30) | 3.0 (2.68) | 8.1 (7.32)
  Year 2 (N: 21, 25) | 8.8 (6.63) | 13.7 (10.51)
  Year 3 (N: 16, 14) | 13.4 (11.31) | 22.3 (11.74)
  Year 4 (N: 8, 7) | 18.6 (17.65) | 36.4 (22.50)
  Year 5 (N: 2, 2) | 30.5 (21.92) | 46.5 (34.65)
  Years 1 - 5 cumulatively (N: 33, 36) | 4.3 (3.58) | 8.6 (7.12)

4. Secondary Outcome: Colorectal Polyp Burden
Description: The polyp burden was defined as the sum of the largest diameters of all polyps (>2 mm in size) over Years 1 - 5 cumulatively.
  Weighted colorectal polyp burden over Years 1 - 5 cumulatively was defined as the polyp burden over Years 1 - 5 divided by the number of colonoscopies that the participant had during the study.
Time Frame: Years 1 - 5
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 55 | 51
mm
  Year 1 (N: 27, 30) | 4.0 (1.97) | 4.2 (2.05)
  Year 2 (N: 21, 25) | 6.9 (2.28) | 8.1 (4.06)
  Year 3 (N: 16, 14) | 9.6 (3.14) | 11.6 (4.05)
  Year 4 (N: 8, 7) | 12.9 (3.31) | 18.7 (5.88)
  Year 5 (N: 2, 2) | 20.0 (7.07) | 20.0 (4.24)
  Year 1 - 5 cumulatively (N: 33, 36) | 4.1 (1.68) | 4.3 (1.61)

ADVERSE EVENTS:
Time Frame: Events were reported from randomization through and including 30 calendar days after the last administration of the study drug.
Description: The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Celecoxib | Placebo
Serious Adverse Events (participants affected / at risk) | 3/53 | 0/48
Other Adverse Events (participants affected / at risk) | 36/53 | 30/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Celecoxib (N=53) | Placebo (N=48)
Periorbital cellulitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Celecoxib (N=53) | Placebo (N=48)
Abdominal discomfort (Gastrointestinal disorders) | 9 | 4
Abdominal pain (Gastrointestinal disorders) | 9 | 10
Abdominal pain upper (Gastrointestinal disorders) | 4 | 3
Diarrhoea (Gastrointestinal disorders) | 6 | 4
Nausea (Gastrointestinal disorders) | 8 | 8
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 3
Vomiting (Gastrointestinal disorders) | 9 | 9
Chest pain (General disorders) | 4 | 1
Fatigue (General disorders) | 6 | 4
Seasonal allergy (Immune system disorders) | 2 | 5
Ear infection (Infections and infestations) | 4 | 2
Gastroenteritis (Infections and infestations) | 3 | 2
Gastroenteritis viral (Infections and infestations) | 3 | 1
Influenza (Infections and infestations) | 6 | 1
Nasopharyngitis (Infections and infestations) | 6 | 4
Upper respiratory tract infection (Infections and infestations) | 4 | 9
Viral infection (Infections and infestations) | 0 | 4
Albumin urine present (Investigations) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 5
Headache (Nervous system disorders) | 16 | 14
Migraine (Nervous system disorders) | 2 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 5

LIMITATIONS AND CAVEATS:
The study was early terminated and, due to the low number of participants, no efficacy analysis was performed. Only descriptive statistics was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.